CLINICAL TRIAL: NCT04149990
Title: Angiotensin-Neprilysin Inhibition in Diastolic Dysfunction After AMI
Acronym: ARNiAMI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Jacob Moller (Other)
Collaborators: Danish Heart Foundation (Other); Odense University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jacob Moller, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Version 1.4
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Infarction; Diastolic Dysfunction
MeSH Terms: conditions — Myocardial Infarction | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Entresto (Active Comparator): Combination of valsartan and sacubitril titrated to 103+97 mg B.I.D. for 26 weeks
  Interventions: Drug: Entresto Pill
- Placebo (Placebo Comparator): Matching placebo B.I.D. for 26 weeks
  Interventions: Drug: Entresto Pill

INTERVENTIONS:
Drug: Entresto Pill — NO other interventions
  Other Names: Valsartan+ sacubitril

SUMMARY:
This study examines the effect of Entresto on central hemodynamic parameters during exercise in patients with diastolic dysfunction following acute myocardial infarction. Half of the patients will receive Entresto and the other half will receive placebo.

DETAILED DESCRIPTION:
In patients with acute myocardial infraction (AMI) only 25-33% have entirely normal left ventricular (LV) systolic and diastolic function. Studies have show that echocardiographic signs of increased LV filling pressure (diastolic dysfunction) are associated with poor outcome after AMI. The optimal management of this group of patients is currently not known. LCZ696 is a novel combination drug consisting of two antihypertensives, sacubitril and valsartan. LCZ696 have demonstrated to reduce mortality in patients with systolic heart failure. In patients with heart failure with preserved ejection fraction a positive effect has been demonstrated on natriuretic peptides and left atrial remodelling when treated with LCZ696, further, experimental data suggest inhibition of cardiac fibrosis.

Hypothesis:

LCZ696 compared with placebo will improve central hemodynamics (reduce pulmonary capillary wedge pressure (PCWP)), and increase cardiac index (CI) during exercise in patients with diastolic dysfunction following AMI. A beneficial effect that is attributed to improved cardiac remodelling (attenuation of cardiac fibrosis).

Primary objective To asses the effect of 6 months treatment with LCZ696 compared with placebo on ratio of PCWP/CI during exercise in patients with a recent AMI and Doppler echocardiographic signs of diastolic dysfunction and preserved systolic function.

ELIGIBILITY:
Inclusion Criteria:

1. Documented ST segment elevation or non ST- myocardial infarction according to current guidelines
2. Complete revascularization
3. Age ≥50 years
4. LVEF ≥45% on echocardiography performed within 72 hours of the MI.
5. Diastolic dysfunction defined as: Ratio of early diastolic peak mitral inflow velocity (E) to early mitral annulus diastolic velocity (e') ratio > 8 and at least moderate LA dilatation (LA volume index>34 mL/m2).
6. Signed informed consent

Exclusion Criteria:

1. Intolerance towards study medication
2. Permanent atrial fibrillation,
3. Known history of cardiomyopathy,
4. More than mild valvular heart disease,
5. Severe obstructive or restrictive pulmonary disease,
6. Inability to perform exercise testing,
7. Inadequate acoustic windows on echocardiography,
8. Ongoing treatment with an angiotensin converting enzyme inhibitor at randomization.
9. Class I indication for an angiotensin converting enzyme inhibitor
10. Symptomatic hypotension, a systolic blood pressure of less than 100 mm Hg at screening
11. An estimated glomerular filtration rate (eGFR) below 30 ml per minute per 1.73 m2 of body-surface area at any time,
12. A serum potassium level of more than 5.2 mmol per liter at screening,
13. A history of hereditary or idiopathic angioedema or unacceptable side effects during receipt of angiotensin converting enzyme inhibitor or angiotensin receptor blocker
14. Inability to provide informed consent
15. Concomitant use of drugs containing aliskiren in patients with diabetes mellitus.
16. Severe reduced liver function, biliary cirrhosis or cholestasis (Child-Pugh class C)
17. Pregnant or nursing(lactating) women(see section 8.2.1 for details)
18. Fertile women unless they are using a highly effective method of contraception(see section 8.2.2 for details)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Central hemodynamics | 26 weeks
  The primary endpoint will be the ratio of mean PCWP at peak exercise divided by cardiac index at peak exercise.

SECONDARY OUTCOMES:
cardiac MRI | 26 weeks
  Amount of hyperenhancement on cardiac MRI using a semiquantitative assessment of late gadolinium hyperenhancement in a 17 segment model of the LV.
Biomarker 1 | 26 weeks
  ST2 concentration at rest.
Biomarker 2 | 26 weeks
  MR-proANP at rest.
Biomarker 3 | 26 weeks
  NT-proBNP at rest.
Echocardiographic 1 | 26 weeks
  Left atrial volume by echocardiography and left atrial emptying fraction by echocardiography at rest.
Echocardiographic 2 | 26 weeks
  Proportion of patients with moderate or severe diastolic dysfunction at rest.echocardiography at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hartmund Frederiksen, DMSC, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Department of Cardiology, Rigshospitalet, Copenhagen
  - Department of Cardiology, Odense Universityhospital, Odense

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04149990/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT04149990/SAP_001.pdf